CLINICAL TRIAL: NCT06624371
Title: Atovaquone Combined With Radiation in Children With Malignant Brain Tumors
Acronym: AflacBT2303
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Morningside Foundation/Peach Bowl LegACy Fund (Unknown)
Responsible Party: Principal Investigator, Tobey MacDonald, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007693
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: High-grade Glioma; Medulloblastoma; Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: Atovaquone; Progression-free survival
MeSH Terms: conditions — Glioma; Medulloblastoma; Diffuse Intrinsic Pontine Glioma | interventions — Atovaquone; Radiotherapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: In Stratum 1, six subjects will be enrolled for a Phase I safety evaluation of atovaquone with radiotherapy (RT). Patients will take atovaquone orally once daily for at least 7 days and up to 21 days before starting RT, continuing through RT without interruption. The study will use a Rolling-6 design with no dose escalation. If no more than one dose-limiting toxicity (DLT) or drug discontinuation for over two weeks due to intolerance occurs in the first six subjects, six additional patients will be enrolled to confirm the safety of the combination. If two or more DLTs or unique drug discontinuations are observed among these twelve patients, the regimen will be deemed too toxic.
  In Stratum 2, six subjects will receive atovaquone daily for six months. Given prior safety in pediatric patients, DLTs are not expected. However, if two or more DLTs or prolonged discontinuations occur, the regimen will also be considered too toxic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stratum 1: (Experimental): Newly diagnosed pHGG/DMG/DIPG patients.
  New Diagnosis followed by 2 weeks (+/- 7 days) atovaquone followed by approx. 6 weeks Atovaquone + Radiotherapy
  Interventions: Drug: Atovaquone; Radiation: Radiation Therapy
- Stratum 2 (Experimental): Stratum 2 will be bifurcated into:
  * Stratum 2a (patients with relapse or progression)
  * Stratum 2b (patients without progression after radiation)
  The same dosing regimen for atovaquone will be used for up to 6 months in the absence of toxicity, intolerance, or tumor progression. Patients will begin therapy between 2-4 weeks after documented relapse or progression of tumor or between 2-4 weeks after completion of standard RT for pHGG/DMG/DIPG patients who have completed standard Radiotherapy without previous atovaquone treatment.
  Interventions: Drug: Atovaquone; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Atovaquone — Atovaquone oral suspension (750 mg/5mL) will be administered with meals on an outpatient basis.
  Patients 13 years and older will receive atovaquone 750 mg PO BID, the standard pediatric dosing for Pneumocystis Jirovecii Pneumonia (PJP) prevention and treatment.
  For those aged 2-12 years, atovaquone will be dosed at 30mg/kg once daily. The maximum dose for children under 12 will be 1500 mg.
Radiation: Radiation Therapy — 54-60 Gy in 1.8 Gy daily fractions of MRI-guided proton radiotherapy using intensity-modulated pencil-beam scanning technology to match the target will be used.
  Other Names: Standard of Care

SUMMARY:
The goal of this interventional study is to Assess the safety and tolerability of atovaquone in combination with standard radiation therapy (RT) for the treatment of pediatric patients with newly diagnosed pediatric high-grade glioma/diffuse midline glioma/diffuse intrinsic pontine glioma (pHGG/DMG/DIPG).

The secondary aim is to assess the safety and tolerability of longer-term atovaquone treatment for pediatric patients with relapsed or progressed pHGG/DMG/DIPG and medulloblastoma (MB) or pHGG/DMG/DIPG after completion of RT and before progression.

DETAILED DESCRIPTION:
Atovaquone, an FDA-approved antiparasitic drug, is being explored as a potential treatment for certain cancers, particularly leukemia and pediatric brain tumors like high-grade gliomas. Since Atovaquone's safety and dosage are already established, repurposing it for cancer treatment is cost-effective.

Research shows that Atovaquone can inhibit a protein called STAT3, which is involved in cancer cell survival and immune response suppression. By doing this, it may enhance the effectiveness of radiation therapy, especially in tumors with low oxygen levels. In animal studies and early clinical trials, Atovaquone has shown promise in reducing tumor size and improving survival rates.

For pediatric brain tumors, which often resist standard treatments, Atovaquone's ability to cross the blood-brain barrier could make it particularly valuable. Ongoing clinical trials are examining its effects in combination with radiation therapy for treating newly diagnosed high-grade gliomas and relapsed medulloblastomas. Overall, Atovaquone's repurposing could lead to new, effective treatment options for difficult-to-treat cancers in children.

ELIGIBILITY:
Inclusion Criteria:

-Stratum 1

* Newly diagnosed pHGG/DMG/DIPG Patients must have histologically confirmed pediatric high-grade glioma (pHGG, WHO Grade 3 or 4) or diffuse midline glioma with altered H3K27 (DMG, WHO Grade 4). Primary pHGG or DMG spinal tumors are eligible. Diffuse intrinsic pontine glioma (DIPG) defined by MRI does not require histological confirmation.
* Weight > 10kg
* Karnofsky and Lansky performance score > 50%
* Patients with stable seizures (e.g., no seizures for ≥ 7 days and not requiring escalation or addition of anti-epileptic drugs) will be eligible.
* Adequate liver function defined as:

  * Total bilirubin ≤ 2x upper limit of normal (ULN) and
  * AST (SGOT) and ALT (SGPT) ≤ 225 U/L (5x the ULN). The ULN for AST and ALT will be 45 U/L.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count > 1,000/mcL
  * platelets > 100,000/mcL
  * hemoglobin > 8g/dL
  * Total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) < 5 x (<10 x if taking steroids) the institutional upper limit of normal
  * creatinine within normal institutional limits for age 2 OR
  * creatinine clearance > 60mL/min/1.73 m for patients with creatinine levels above institutional normal

Stratum 2

* Relapsed, progressive pHGG/DMG/DIPG and medulloblastoma (MB) or pHGG/DMG/DIPG after completion of standard radiation therapy without prior atovaquone exposure and before progression. Patients with metastatic disease are allowed for Stratum 2 only.

  --Measurable disease is not necessary for enrollment study.
* Patients must have previously undergone standard-of-care treatment including surgery, radiation, and/or first-line adjuvant chemotherapy before the experimental treatment (atovaquone).
* Patients must have recovered from the acute treatment-related toxicities (defined as < grade 1 if not defined in eligibility criteria) of all prior chemotherapy, immunotherapy or radiotherapy prior to entering this study. There is no upper limit to the number of prior therapies that is allowed.
* Age > 2 to 25 years
* Weight > 10kg
* Karnofsky and Lansky performance score > 50%
* Patients with stable seizures (e.g., no seizures for ≥ 7 days and not requiring escalation or addition of anti-epileptic drugs) will be eligible.
* Patients must have normal organ and marrow function as defined above for Stratum 1
* Adequate liver function is defined as:

  1. Total bilirubin ≤ 2x upper limit of normal (ULN) and
  2. AST (SGOT) and ALT (SGPT) ≤ 225 U/L (5x the ULN). The ULN for AST and ALT will be 45 U/L.

Exclusion Criteria:

Stratum 1

* Chronic systemic concurrent illness
* Concurrent or history of anti-cancer therapy other than RT
* Patients with metastatic tumor are excluded for Stratum 1 only.
* Patients with uncontrolled seizures or seizure requiring escalation or addition of anti-epileptic drugs are excluded.
* Patients must fully recover from all acute effects of prior surgical intervention.
* History of allergic reactions to atovaquone or attributed to compounds of similar chemical or biological composition to atovaquone.
* Symptomatic intratumoral hemorrhage, or asymptomatic intratumoral hemorrhage larger than punctate foci, at any time prior to enrollment.
* Pregnant or breast-feeding women will not be entered into this study as there may be fetal risks or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during treatment and for 3 months after stopping treatment. This should be documented in the electronic medical records as part of the consent discussion.

Stratum 2

* Concurrent illness
* Patients must have recovered from all prior therapy as follows:

  1. Patients must have received their last dose of known myelosuppressive anticancer therapy at least three (3) weeks before study enrollment or at least six (6) weeks if prior nitrosourea.
  2. Biologic or investigational agent (anti-neoplastic): Patient must have received their last dose of the investigational or biologic agent ≥ 7 days before study enrollment.
  3. Antibodies: ≥ 21 days must have elapsed from an infusion of the last dose of antibody and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1. Agents with prolonged half-lives: At least three half-lives must have elapsed before enrollment.
  4. Immunotherapy: Patient must have completed immunotherapy (e.g. tumor vaccines, oncolytic viruses. etc.) at least 42 days before enrollment.
  5. Radiation: Patients must have had their last fraction of • Craniospinal irradiation ≥ 3 months before enrollment. • Other substantial bone marrow irradiation ≥ 6 weeks before enrollment • Local or palliative XRT (small port) ≥ 2 weeks.
  6. Stem Cell Transplant: Patient must be ≥ 12 weeks since autologous bone marrow/stem cell transplant before enrollment. Patients with uncontrolled seizures or seizure requiring escalation or addition of anti-epileptic drugs are excluded.
* Patients must fully recover from all acute effects of prior surgical intervention.
* History of allergic reactions to atovaquone or attributed to compounds of similar chemical or biological composition to atovaquone.
* Pregnant or breast-feeding women will not be entered into this study as there may be fetal risks or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during treatment and for 3 months after stopping treatment. This should be documented in the electronic medical records as part of the consent discussion.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Drug Limiting toxicities (DLT) in Stratum 1 | Baseline, end of study (10 weeks)
  Adverse events that meet definition of DLT and tolerability. The outcome will be evaluated by descriptive statistics. Rates of symptomatic and asymptomatic radiation necrosis will also be estimated for Stratum 1 patients.
Drug Limiting toxicities (DLT) in Stratum 2 | Baseline, End of study (Month 7)
  Adverse events that meet definition of DLT and tolerability. The outcome will be evaluated by descriptive statistics. Rates of symptomatic and asymptomatic radiation necrosis will also be estimated for Stratum 2 patients.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) in newly diagnosed pediatric high-grade glioma/diffuse midline glioma/diffuse intrinsic pontine glioma (pHGG/DMG/DIPG) patients (Stratum 1) | Baseline, Month 12
  PFS is defined as the time from initiation of drug treatment to the occurrence of confirmed disease progression. Subjects who are lost to follow-up or withdraw from the study will be treated as censored observations at the last follow-up time point when they are alive.
Progression Free Survival (PFS) in Stratum 2 subjects | Baseline, Month 12
  PFS is defined as the time from initiation of drug treatment to the occurrence of confirmed disease progression. Subjects that are lost to follow-up or withdraw from the study will be treated as censored observations at the last follow-up time point when they are alive.
Overall survival (OS) in newly diagnosed pHGG/DMG/DIPG patients (Stratum 1) | Baseline, end of study (Week 10)
  OS is defined as time from enrollment to death due to any cause. The Kaplan-Meier method will be used to estimate the OS rates over time. Median survival time along with 95% confidence interval (CI) will be calculated
Overall survival in Stratum 2 subjects | Baseline, End of study (Month 7)
  OS is defined as time from enrollment to death due to any cause. The Kaplan-Meier method will be used to estimate the OS rates over time. Median survival time along with 95% confidence interval (CI) will be calculated
Objective Tumor Response Rate (ORR) for Stratum 2 | Baseline, End of study (Month 7)
  Objective response (PR or CR), observed anytime during treatment and sustained for at least 8 weeks, in patients with relapsed or progressive pHGG, DMG/DIPG, or MB.
  Complete Response (CR): Complete disappearance on MR of all evaluable tumor and mass effect, on a stable or decreasing dose of corticosteroids (or receiving only adrenal replacement doses),accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks.
  If CSF was positive, it must be negative. Partial Response (PR): Greater than or equal to 50% reduction in tumor size by bi-dimensional measurement, as compared with the baseline measurements, on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Tobey MacDonald, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Arthur M Blank Hospital, Atlanta, Georgia
  - Children's Healthcare of Atlanta: Scottish Rite, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No